CLINICAL TRIAL: NCT03723330
Title: Impact of Co-consuming a Plant Sterols-enriched Food Product With a Healthy Eating Pattern Diet on Endothelial Function and Blood Pressure Management in Individuals With Metabolic Syndrome
Brief Title: Impact of Consuming Plant Sterols on Endothelial Function and Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Jung Eun Kim, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: S6
Record Dates: First submitted 2018-10-23; First posted 2018-10-29 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Cardiovascular Diseases; Endothelial Dysfunction; Metabolic Syndrome; Diet Modification
Keywords: Endothelial function; Blood pressure; healthy diet
MeSH Terms: conditions — Cardiovascular Diseases; Metabolic Syndrome | interventions — Phytosterols; Diet, Healthy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plant sterol with a healthy diet (Experimental): Each subject will be provided one-to-one dietary counselling by a research dietitian and an instruction sheet to achieve the healthy eating pattern diet. Subjects will also be provided with specific instructions to consume plant sterols-enriched food (contains 2 g plant sterols).
  Interventions: Dietary Supplement: plant sterols; Other: healthy diet
- Healthy diet (Active Comparator): Each subject will be provided one-to-one dietary counselling by a research dietitian and an instruction sheet to achieve the healthy eating pattern diet.
  Interventions: Other: healthy diet

INTERVENTIONS:
Dietary Supplement: plant sterols — Consumption a healthy eating pattern diet with a plant sterols-enriched food product
  Arms: Plant sterol with a healthy diet
Other: healthy diet — Compliance with a healthy diet in accordance to the recommendation by the Singapore Health Promotion Board.

SUMMARY:
The purpose of the research is to assess the impact of co-consuming plant sterols-enriched food product as part of a healthy eating pattern diet on endothelial function (brachial artery FMD, vasodilation-related and vasoconstriction-related biomarkers) and blood pressure management (24-hour ambulatory and classic blood pressure) in Singapore individuals with MetS.

DETAILED DESCRIPTION:
This is a 13-wk double-blinded, randomized, crossover study design. Following a 1-wk pre-intervention baseline period, subjects will be randomly assigned to follow a healthy eating pattern diet either contain 2.0 g free plant sterols equivalent of their palmityl esters (Plant Sterol Diet) or do not contain plant sterols (Control Diet) for 4 weeks. After a 4-week dietary 'washout' period, they will consume the alternative diet for 4 weeks. The random assignment will be done with SAS 9.4 software. Body size measurement, dietary assessment, brachial artery FMD and blood pressure measurements, and fasting-state blood collection will be conducted at week 1, 5, 9, and 13, which correspond to before and during the last 1 week of the two 4-week intervention periods.

During study week 1 and weeks 6-9, all subjects will consume their habitual, unrestricted self-chosen diets. During study weeks 2-5 and 10-13, all subject will follow a healthy eating pattern diet, referred to as the "My Healthy Plate" designed by HPB. Each subject's energy requirement will be estimated using sex-specific equations and Recommended Dietary Allowances for healthy Singaporean. One-on-one dietary counselling and written instructions for each subject will be provided by a research dietitian and trained research staff to achieve a healthy eating pattern diet. Compliance with the plant sterols consumption will be promoted by frequent online and in-person contact.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to give an informed consent;
2. Age>35 years old;
3. Meet any 3 of the 5 following NCEP-ATP III MetS criteria (waist circumference > 90 cm (male), > 80 cm (female); fasting glucose concentration ≥ 100 mg/dL or on medication; triglyceride ≥ 150 mg/dL or on medication; high density lipoprotein cholesterol (HDL) < 40 mg/dL (male), < 50 mg/dL (female); systolic or diastolic blood pressure > 130/80 mmHg or on medication);
4. Weight change < 3kg in the past 3 months;
5. No exercising vigorously over the past 3 months;
6. No allergy to plant sterols; no acute illness; not smoking;
7. No drinking more than 2 alcoholic drinks per day;
8. No pregnant, lactating, or planning pregnancy in the next 6 months.

Exclusion Criteria:

1. Unable to give an informed consent;
2. Age<35 years old;
3. Meet less than 3 of following NCEP-ATP III MetS criteria (waist circumference > 90 cm (male), > 80 cm (female); fasting glucose concentration ≥ 100 mg/dL or on medication; triglyceride ≥ 150 mg/dL or on medication; high density lipoprotein cholesterol (HDL) < 40 mg/dL (male), < 50 mg/dL (female); systolic or diastolic blood pressure > 130/80 mmHg or on medication);
4. Weight change > 3kg in the past 3 months;
5. Exercise vigorously over the past 3 months;
6. Allergy to plant sterols; no acute illness; not smoking;
7. Drinking more than 2 alcoholic drinks per day;
8. Pregnant, lactate, or plan pregnancy in the next 6 months.

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Change in brachial artery flow-mediated dilation (FMD) | Every 4 weeks (Week 1, week 5, week 9, week 13)
  Brachial artery FMD will be measured by high-frequency and ultrasonographic imaging.
Change in vasodilation and vasoconstriction related biomarkers | Every 4 weeks (Week 1, week 5, week 9, week 13)
  Vasodilation and vasoconstriction related biomarkers contains nitric oxide, endothelial nitric oxide synthase, and endothelin-1. They will be measured using the commercially available ELISA assay kits.
Change in blood pressure | Every 4 weeks (Week 1, week 5, week 9, week 13)
  Classical and 24-hour ambulatory blood pressure: Systolic and diastolic blood pressure and 5-day of 24-hour ambulatory blood pressure will be measured.

SECONDARY OUTCOMES:
Change in blood lipid-lipoproteins | Every 4 weeks (Week 1, week 5, week 9, week 13)
  Assessing the blood lipid-lipoproteins profile includes the measurements of plasma total cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, and triglyceride concentrations.
Change in skin carotenoid status | Every 4 weeks (Week 1, week 5, week 9, week 13)
  Measured using resonance Raman spectroscopy.
Height | Pre-intervention only
  Height (cm)
Change in weight | Every 4 weeks (Week 1, week 5, week 9, week 13)
  Weight (kg)
Change in waist circumference | Every 4 weeks (Week 1, week 5, week 9, week 13)
  Waist circumference (cm)
Change in diet | Every 4 weeks (Week 1, week 5, week 9, week 13)
  Dietary assessment, 3-day food record
Change in sleep quality (Pittsburgh sleep quality index questionnaire (PSQI)) | Every 4 weeks (Week 1, week 5, week 9, week 13)
  Recall based questionnaire assessing sleep habits for the past one month only which includes sleeping timing habits and quality of sleep (Very good, Fairly good, Fairly bad and very bad)

CONTACTS AND LOCATIONS:
Overall Officials: J Eun Kim, PhD, Principal Investigator — National University of Singapore
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Electronic copies of the data with identifiable participant information will be kept, data will be de-identified prior to be statistical analysis.

REFERENCES:
- [Background] Ho XL, Loke WM. Dietary Plant Sterols Supplementation Increases In Vivo Nitrite and Nitrate Production in Healthy Adults: A Randomized, Controlled Study. J Food Sci. 2017 Jul;82(7):1750-1756. doi: 10.1111/1750-3841.13752. PMID 28708316
- [Derived] Xu Y, Sutanto CN, Xia X, Toh DWK, Gan AX, Deng Q, Ling LH, Khoo CM, Foo RS, Kim JE. Consumption of plant sterols-enriched soy milk with a healthy dietary pattern diet lowers blood pressure in adults with metabolic syndrome: A randomized controlled trial. Nutr Metab Cardiovasc Dis. 2025 Jan;35(1):103773. doi: 10.1016/j.numecd.2024.10.011. Epub 2024 Oct 16. PMID 39561689